CLINICAL TRIAL: NCT05296993
Title: The Safety and Effectiveness of the Extended Longevity Protocol on the Epigenetic Aging Rate in Healthy Individuals
Brief Title: Safety & Efficacy of Extended Longevity Protocol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TD-EL-001
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracts (Experimental): The ingredients found in these serums are all naturally occurring ingredients extracted from a variety of plant species: Pinetonal, Thyvolve, Telogenic, Sentophagy, Inflasolve, Stemegenis, and CMEnhance
  Interventions: Dietary Supplement: Extracts found in the Extended Longevity supplements

INTERVENTIONS:
Dietary Supplement: Extracts found in the Extended Longevity supplements — Ingredients found in these serums are all naturally occurring, and extracted from a variety of plant species.

SUMMARY:
The purpose of this study is to quantifiably determine if the Extended Longevity Protocol has a significant clinical effect on epigenetic age.

DETAILED DESCRIPTION:
This is a prospective non-randomized clinical study of 15 patients to determine if the safety and effectiveness of the Extended Longevity Protocol's impact on the nine determinant factors of aging can decelerate aging.

There is evidence that the Extended Longevity Protocol decelerates aging and the risk of age-related diseases. The aim of this pilot study is to evaluate the safety, efficacy and feasibility of the Extended Longevity Protocol as an effective treatment option to improve clinical care of healthy individual's biological age thus prolonging longevity.

ELIGIBILITY:
Inclusion Criteria:

* 8 Men and 7 Women
* Must between 55-75 years old
* Patient must be able to comply with treatment plan and laboratory tests
* Patients must have adequate immune system function, with no known immunodeficiency disease

Exclusion Criteria:

* Neoplastic cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
* No immune system issues or immunodeficiency disease
* No history of viral illness which could be reactivated by immune downregulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke) disease
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Patients infected with hepatitis, C or HIV
* Patients with Body Mass Index (BMI) > 40 kg/m2
* Presence of active infection
* Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the investigator would render a patient unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age | Testing will compare the change in results from baseline to 3 months
  Serum epigenetic aging test
Epigenetic Age | Testing will compare the change in results after completion of intervention with baseline
  serum epigenetic aging test

CONTACTS AND LOCATIONS:
Locations (1):
- Quantum Functional Medicine, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: Undecided